CLINICAL TRIAL: NCT05773820
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of WJB001 Capsules in Dose Escalation, Dose Expansion, and Efficacy Expansion in Patients With Advanced Solid Tumors
Brief Title: A Study Explore WJB001 Capsules in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wigen Biomedicine Technology (Shanghai) Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WJB001-001-I
Record Dates: First submitted 2023-02-16; First posted 2023-03-17 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WJB001 capsules (Experimental): Once a day (QD).
  Interventions: Drug: WJB001

INTERVENTIONS:
Drug: WJB001 — Dose Escalation:
  Accelerated titration (the first two dose groups) and "BOIN" combination (the subsequent dose group) were used for dose escalation.
  Dose Expansion:
  Based on the previous data, 1 to 2 doses were selected to further evaluate the initial efficacy, safety, tolerability and pharmacokinetic characteristics to confirm RP2D.
  Cohort Expansion:
  The preliminary plan of cohort expansion phase uses the Simon two-stage optimal method to expand 2 to 3 cohorts.

SUMMARY:
This is a phase I/II study to evaluate the safety and tolerability, DLT(Dose limited toxicity), MTD(Maximum tolerated dose), and RP2D(Recommended phase II dose) of WJB001 capsules in patients with advanced solid tumors, including dose escalation phase, dose expansion phase and cohort expansion phase.The study includes screening, treatment and follow-up periods.

In the Dose Escalation phase:Accelerated titration (the first two dose groups) and "BOIN" combination (the subsequent dose group) were used for dose escalation.

In the Dose Expansion phase:Based on the previous data, 1 to 2 doses were selected to further evaluate the initial efficacy, safety, tolerability and pharmacokinetic characteristics to confirm RP2D.

In the Cohort Expansion phase:The preliminary plan of cohort expansion phase uses the Simon two-stage optimal method to expand 2 to 3 cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

1. ≥ 18 years or older at the time of informed consent；
2. Patient with advanced malignant solid tumors clearly diagnosed pathologically and/or cytologically, who have failed to receive standard treatment, or who currently no have standard treatment, or who are intolerant to standard treatment;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score ≤1;
4. Life expectancy ≥ 12 weeks;
5. Adequate hematologic and organ function；
6. All acute toxic effects from previous antineoplastic therapy or surgery ；
7. Fertile women must confirm a negative blood pregnancy test within 7 days prior to the first administration of study drug;and they required to use adequate and effective contraceptive measures throughout the treatment period and within 3 months after the end of treatment;Fertile women in this protocol were defined as sexually mature women: 1) not undergoing hysterectomy or bilateral oophorectomy; 2) 24 months without a continuous period of spontaneous menopause (i.e., having had a period at any time in the previous 24 consecutive months; Amenorrhea after cancer treatment does not exclude fertility). Male participants with a sexual partner who was a woman of reproductive age had to agree to use an effective contraceptive method while using the study drug and for 3 months after the last dose；

   Specific inclusion criteria：
8. At least one measurable tumor lesion that meets the definition of RECIST v1.1, with no history of biopsy two weeks before screening(applicable to all stages);
9. Subjects with CCNE1 overexpression (H score > 50) or amplification (DNA copy number > 7)confirmed by central laboratory (applicable to the dose expansion stage and efficacy expansion stage);
10. For subjects with advanced uterine serous carcinoma, ≤2 lines of therapy for recurrence are allowed after first-line treatment; For subjects with advanced high-grade serous ovarian, fallopian tube, or peritoneal cancer,≤2 lines of therapy after platinum resistance are allowed(applicable to the dose expansion stage and efficacy expansion stage)；

Key Exclusion criteria：

1.General condition

1. Pregnant or lactating women;
2. Any known allergies to or contraindications to components of the study drug;
3. History of substance abuse;
4. History of alcohol abuse or consumption of more than 28 units of alcohol per week (1 unit =285 ml beer or 25 ml spirits (40%v/v) or 100 ml wine).

2.Previous or current treatment:

1. Previous or current treatment with Wee1 inhibitors;
2. Received cytotoxic chemotherapy drugs,anti-tumor traditional Chinese medicine orother anti-tumor therapies (such as small molecule targeted therapy, etc.)within 4 weeks prior to the first administration of study drug;Or received the investigational drug, macromolecular drug with anti-tumor effect (e.g., monoclonal antibody, antibody-drug conjugate, or bispecific antibody, etc.) within 28 days prior to the first administration of study drug; Or need to continue receiving these medications during the study;
3. The use of a medium or strong inhibitor or inducer of CYP3A or other product (e.g., grapefruit juice) or P-gp inhibitor or inducer was discontinued less than the time before the first dose of WJB001 was administered 5 half-lives of the drug or 14 days, whichever is shorter;
4. Patients with a known organ transplant or stem cell transplant; Major surgery or major trauma (excluding needle biopsy for sample collection) within 4 weeks prior to the first administration of study drug;
5. Radiation therapy was administered within 21 days prior to the first administration of study drug; (except the radiation was delivered to ≤5% of bone marrow volume).3. Past medical history, present medical history and abnormal laboratory indicators:

3. Abnormal laboratory indicators:

1. Having active GI abnormalities including, but not limited to, inability to take oral medication, need for intravenous nutritional support, peptic ulcer, chronic diarrhea (e.g., Crohn's disease, irritable bowel syndrome), or vomiting or other factors that the investigator believes may significantly affect drug absorption, metabolism, or excretion;
2. History of severe ocular disease (except permanent blindness due to disease) that has not recovered to grade 1 or less;
3. Patients with active brain metastases (except if they had CNS metastases confined to the supratentorial or cerebellar region, had been adequately treated (surgery or radiotherapy), had maintained radiological stability for at least 4 weeks, and did not require corticosteroids for symptom control);
4. Patients with current cancer meningitis or spinal cord compression;
5. Severe or poorly controlled hypertension, including previous history of hypertensive crisis or hypertensive encephalopathy; Adjustment of antihypertensive medication due to poor blood pressure control within 2 weeks before the first dose;Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg during the screening period;
6. Patients with clinically significant bleeding symptoms or obvious bleeding tendency within 4 weeks before the first dose, such as gastrointestinal bleeding, gastric ulcer bleeding, obvious gross hematuria, or angiitis;
7. Patients with active HBV and HCV infection: if HBsAg is positive or/and anti-HBc is positive, blood HBV DNA should be tested to confirm that it is above the limit of quantitative detection; If anti-HCV is positive, it is necessary to detect HCV RNA to confirm that the HCV virus copy number exceeds the quantitative detection limit；
8. Known history of human immunodeficiency virus infection or seropositivity for HIV;
9. History of syphilis (both treponema pallidum specific and non-specific antibodies were positive)；
10. History of other primary solid tumor (except a cured solid tumor that has been inactive for ≥5 years before screening and has a very low risk of recurrence）; Adequately treated non-melanoma skin cancer or lentigo maligna with no evidence of disease recurrence; Adequately treated carcinoma in situ with no evidence of disease recurrence, such as carcinoma in situ of the cervix);
11. history of severe or what the investigators considered clinically significant cardiac disease affected the safety assessment；
12. Severe active infectious diseases or other diseases that seriously affect the safety of the first medication occurred during the screening period;
13. There are other factors that the investigator considers may affect the results of the study and interfere with the patient's participation in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
1.Dose limited toxicity (DLT) | 3 years
  incidence of Dose limited toxicity(DLT);
2.Adverse event (AE) | 3 years
  incidence and severity of adverse event (AE), Abnormal changes in laboratory and other tests of clinical significance;
3.Serious adverse event (SAE) | 3 years
  incidence and severity of Serious adverse event (SAE);
4.Maximum tolerated dose (MTD) | 2 years
  Maximum tolerated dose (MTD)
5.Recommended phase II dose (RP2D) | 2 years
  Recommended phase II dose (RP2D)
6.Objective response rate(ORR) | 3 years
  Efficacy endpoints: Objective response rate(ORR) per RECIST v1.1

SECONDARY OUTCOMES:
7. Peak time(Tmax) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Peak time(Tmax) after a single dose;
8.Maximum plasma concentration (Cmax) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Maximum plasma concentration (Cmax) after a single dose;
9. (AUC 0-t) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Area under blood concentration - time curve(AUC 0-t) after a single dose;
10. (AUC 0-∞) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Area under blood concentration - time curve(AUC 0-∞) after a single dose;
11.Apparent volume of distribution (Vd/F) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Apparent volume of distribution (Vd/F) after a single dose;
12.Clearance rate (CL/F) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Clearance rate (CL/F) after a single dose;
13. Elimination half-life time ( t1/2) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Elimination half-life time ( t1/2)
14.Steady state peak concentration(Cmax,ss) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Steady state peak concentration(Cmax,ss) after repeated administration;
15.Steady state valley concentration(Cmin,ss) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Steady state valley concentration(Cmin,ss) after repeated administration;
16.Average steady-state plasma concentration(Cav,ss) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Average steady-state plasma concentration(Cav,ss) after repeated administration;
17. Steady state peak time(Tmax,ss) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Steady state peak time(Tmax,ss) after repeated administration;
18.Steady state Area under blood concentration - time curve(AUC0-t,ss) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Steady state Area under blood concentration - time curve(AUC0-t,ss) after repeated administration;
19.Accumulation Index ( RAC) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter :Accumulation Index ( RAC) after repeated administration;
20.Fluctuation coefficient (FD) | Prior to dose on day 1,5,8,12 and at 0.5,1,1.5, 2,3, 4, 6,8,10 and 24 hours post dose on day 1 and day 12 of Cycle 1
  Pharmacokinetic (PK) parameter : Fluctuation coefficient (FD)
21.Duration of response (DOR) | 3 years
  Efficacy endpoints: Duration of response (DOR) per RECIST v1.1
22.Disease control rate (DCR) | 3 years
  Efficacy endpoints: Disease control rate (DCR) per RECIST v1.1
23.Progression-free survival (PFS) | 2 years
  Efficacy endpoints: Progression-free survival (PFS) per RECIST v1.1
24. Overall survival (OS) | 3 years
  Efficacy endpoints: Overall survival (OS) per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Professor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (10):
- China (10):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - Henan Cancer Hospital, Henan, Zhenzhou

IPD SHARING:
Plan to Share IPD: No